CLINICAL TRIAL: NCT02775162
Title: A Multicenter Randomized Controlled Trial to Compare the Efficacy of Ex-vivo Normothermic Machine Perfusion With Static Cold Storage in Human Liver Transplantation
Brief Title: WP01 - Normothermic Liver Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrganOx Ltd. (Industry)
Collaborators: North American Science Associates Ltd. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WP01
Record Dates: First submitted 2016-03-30; First posted 2016-05-17 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Standard of Care; Ice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normothermic Machine Perfusion (NMP) (Experimental): Following the routine retrieval procedure of the liver, it will be placed on the OrganOx metra for Normothermic Machine Perfusion (NMP) for transport per the Investigational Plan and the Instructions For Use.
  Interventions: Device: Normothermic Machine Perfusion (NMP)
- Standard of Care (Ice) (Other): Following the routine retrieval procedure of the liver, it will be placed in ice-cold perfusion solution within an ice box for transport as dictated by logistics and local policy.
  Interventions: Other: Standard of Care (Ice)

INTERVENTIONS:
Device: Normothermic Machine Perfusion (NMP)
  Other Names: OrganOx metra® device
  Arms: Normothermic Machine Perfusion (NMP)
Other: Standard of Care (Ice)
  Arms: Standard of Care (Ice)

SUMMARY:
A multicenter randomized controlled trial to compare the efficacy of ex-vivo normothermic machine profusion with static cold storage in human liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or greater
* Subject is registered as an active recipient on the United Network for Organ Sharing (UNOS) waiting list for liver transplantation
* Subject, or legally authorized representative, is able and willing to give informed consent and HIPAA authorization
* Subject is able and willing to comply with all study requirements

Exclusion Criteria:

* Subject requiring all of the following at the time of transplantation: oxygen therapy, inotropic support, renal replacement therapy
* Subject has acute/fulminant liver failure
* Subject undergoing simultaneous transplantation of more than one organ
* Subject is pregnant or nursing
* Concurrent enrollment in another clinical trial. Subjects enrolled in clinical trials or registries where only measurements and/or samples are taken (NO TEST DEVICE or TEST DRUG USED) are allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2016-10-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2021-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Knechtle, MD, Principal Investigator — Duke University
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - University of Southern California (USC), Los Angeles, California
  - University of California - Los Angeles (UCLA), Los Angeles, California
  - University of California-San Francisco (UCSF), San Francisco, California
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Ochsner, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kubal C, Mihaylov P, Holden J. Oncologic indications of liver transplantation and deceased donor liver allocation in the United States. Curr Opin Organ Transplant. 2021 Apr 1;26(2):168-175. doi: 10.1097/MOT.0000000000000866. PMID 33650998

RESULTS

PARTICIPANT FLOW:
Groups:
- Normothermic Machine Perfusion (NMP): Following the routine retrieval procedure of the liver, it will be placed on the OrganOx metra for Normothermic Machine Perfusion (NMP) for transport per the Investigational Plan and the Instructions For Use.
  Normothermic Machine Perfusion (NMP)
- Standard of Care (Ice): Following the routine retrieval procedure of the liver, it will be placed in ice-cold perfusion solution within an ice box for transport as dictated by logistics and local policy.
  Standard of Care (Ice)
Period: Overall Study
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Started | 136 | 131
Completed | 122 | 121
Not Completed | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice) | Total
Number analyzed (Participants) | 136 | 131 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (10.5) | 57.2 (10.6) | 57.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 48 | 91
  Male | 93 | 83 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 121 | 118 | 239
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 127 | 119 | 246
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 136 | 131 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Allograft Dysfunction (EAD)
Description: EAD is a binary outcome defined by the presence of one of the following 3 outcomes:
  * Serum bilirubin ≥ 10 mg/dL at day 7 post-transplant
  * International normalized ratio (INR) ≥ 1.6 at day 7 post-transplant
  * Alanine Aminotransferase (ALT) or Aspartate Transaminase (AST) > 2000 IU/L within the first 7 days post-transplant
Time Frame: 7 Days
Population: There was one subject excluded from the primary endpoint analysis as there was only an attempt to transplant a randomized liver. The subject was deemed unable to proceed with the liver transplant and was followed through 30-days post-transplant for adverse event collection only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 136 | 130
percentage of participants | 20.6 [14.5 to 28.5] | 23.7 [17.1 to 31.9]

2. Secondary Outcome: Number of Participants With Primary Non-Function
Description: Primary Non-Function is defined in this study as irreversible graft dysfunction requiring emergency liver replacement during the first 10 days after liver transplantation.
Time Frame: 10 Days
Population: The overall number of participants analyzed reflects participants in each arm who were eligible to be included in the analysis and had complete data.
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 135 | 129
Participants | 1 | 2

3. Secondary Outcome: Number of Participants With Graft Survival
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 127 | 125
Participants | 124 | 122

4. Secondary Outcome: Number of Participants With Subject Survival
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 127 | 125
Participants | 121 | 123

5. Secondary Outcome: Number of Participants With Post-Reperfusion Syndrome
Description: Post-Reperfusion Syndrome is defined in this study as a decrease in mean arterial pressure (MAP) of more than 30% from the baseline value for more than one minute during the first five minutes after reperfusion.
Time Frame: 1 Day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 136 | 130
Participants | 8 | 19

6. Secondary Outcome: Measure Biochemical Liver Function Via Bilirubin
Time Frame: 6 Months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 125 | 125
mg/dL | 0.6 [0.4 to 0.8] | 0.5 [0.4 to 0.7]

7. Secondary Outcome: Measure Biochemical Liver Function Via Gamma-Glutamyl Transferase (GGT)
Time Frame: 6 Months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 72 | 75
IU/L | 38.5 [21.5 to 78.0] | 34.0 [20.0 to 72.0]

8. Secondary Outcome: Measure Biochemical Liver Function Via Alanine Aminotransferase (ALT)
Time Frame: 6 Months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 125 | 125
IU/L | 23.0 [16.0 to 39.0] | 21.0 [16.0 to 32.0]

9. Secondary Outcome: Measure Biochemical Liver Function Via Aspartate Transaminase (AST)
Time Frame: 6 Months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 125 | 125
IU/L | 24.0 [18.0 to 30.0] | 20.0 [16.0 to 26.0]

10. Secondary Outcome: Measure Biochemical Liver Function Via Alkaline Phosphatase (ALP)
Time Frame: 6 Months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 125 | 125
IU/L | 94.0 [72.0 to 137.0] | 92.0 [68.0 to 115.0]

11. Secondary Outcome: Measure Biochemical Liver Function Via International Normalized Ratio (INR)
Description: The international normalized ratio (INR) is a laboratory measurement of how long it takes blood to form a clot. It is calculated using the following formula: INR = (PT [test] / PT [control])^ISI
  INR = international normalized ratio PT [test] = tested prothrombin time PT [control] = control prothrombin time ISI = international sensitivity index
Time Frame: 6 Months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: No Units
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 106 | 98
No Units | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.1]

12. Secondary Outcome: Measure Biochemical Liver Function Via Lactate
Time Frame: Days 1-7
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 102 | 97
mmol/L | 1.4 [1.0 to 2.1] | 1.5 [1.0 to 1.9]

13. Secondary Outcome: Number of Participants With Evidence of Ischemia-Reperfusion Injury Via Comparison of Pre-Reperfusion Biopsies to Post-Reperfusion Biopsies
Description: Overall Degree of Ischemia Reperfusion Injury (IRI) was categorized as:
  * None/Minimal: None or Polymorphonuclear Leukocytes (PMNs) in sinusoidal zone 3 with rare hepatocellular necrosis
  * Mild: Polymorphonuclear Leukocytes (PMNs) in sinusoidal zone 3 with ≥ 1 cluster of necrotic hepatocytes
  * Moderate/Severe: Clusters of hepatocellular necrosis in > 50% of lobules or 60% of parenchyma or panlobular necrosis in > 1 lobule
Time Frame: 1 Day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 133 | 122
Participants
  Pre-Reperfusion: None/Minimal | 123 | 117
  Pre-Reperfusion: Mild | 10 | 5
  Pre-Reperfusion: Moderate/Severe | 0 | 0
  Post-Reperfusion: None/Minimal | 100 | 93
  Post-Reperfusion: Mild | 29 | 24
  Post-Reperfusion: Moderate/Severe | 4 | 5

14. Secondary Outcome: Number of Participants With Biliary Investigations and Biliary Interventions
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 127 | 126
Participants
  Biliary Investigations | 14 | 16
  Biliary Interventions | 12 | 11

15. Secondary Outcome: Number of Livers Randomized But Not Transplanted
Time Frame: 1 Day
Population: The analysis population for this outcome reflects all livers randomized in the study; therefore, the number analyzed is greater than the participants enrolled.
Measure: Count of Units; unit: Livers
Units Other Than Participants: Livers
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 192 | 191
Number analyzed (Livers) | 192 | 191
Livers | 56 | 61

16. Secondary Outcome: Number of Livers That Did Not Experience a Safety Event
Description: Number of livers that did not experience at least one of the following safety events:
  * Early Allograft Dysfunction (EAD)
  * Discard of a Retrieved Liver
  * Primary Non-Function (PNF)
Time Frame: 10 Days
Population: The analysis population for this outcome reflects all livers retrieved in the study; therefore, the number analyzed is greater than the participants enrolled, but less than the total livers randomized. There was one subject where there was only an attempt to transplant a randomized liver as the subject was deemed unable to proceed with the liver transplant.
Measure: Count of Units; unit: Livers
Units Other Than Participants: Livers
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 152 | 140
Number analyzed (Livers) | 152 | 140
Livers | 147 | 137

17. Secondary Outcome: Assessment of the Health Economic Implications Via Length of ICU Stay and Length of Hospital Stay
Time Frame: 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 134 | 127
Days
  Length of ICU Stay | 4.6 (7.5) | 4.2 (6.2)
  Total Length of Hospital Stay | 14.3 (17.1) | 13.3 (18.1)

18. Secondary Outcome: Compare Quality of Life Via the EQ-5D-5L Quality of Life Questionnaire
Description: The EQ-5D-5L Questionnaire is the standard layout for recording an adult person's current self-reported health state. It consists of a standard format for respondents to record their health state according to the EQ-5D-5L descriptive system and the EQ Visual Analog Scale (VAS). EQ-5D-5L index scores range from 0 to 1.0 on a scale where 0 = death and 1.0 = perfect health. EQ-5D-5L is the name of the instrument and is not an acronym.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
Number analyzed (Participants) | 121 | 116
score on a scale | 0.9 (0.1) | 0.8 (0.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the point of enrollment through study exit (12 months for subjects completing the study).
Arm/Group | Normothermic Machine Perfusion (NMP) | Standard of Care (Ice)
All-Cause Mortality (participants affected / at risk) | 10/136 | 4/131
Serious Adverse Events (participants affected / at risk) | 95/136 | 93/131
Other Adverse Events (participants affected / at risk) | 125/136 | 123/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normothermic Machine Perfusion (NMP) (N=136) | Standard of Care (Ice) (N=131)
Chest Infection (Infections and infestations) | 0 | 1
Blood Infection (Infections and infestations) | 11 | 6
Biliary Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Abdominal Infection (Infections and infestations) | 2 | 5
Gastrointestinal Infection (Infections and infestations) | 5 | 3
Skin Infection (Infections and infestations) | 1 | 0
Infection Other (Infections and infestations) | 1 | 3
Bile Leak (Hepatobiliary disorders) | 3 | 4
Biliary Stricture (Anastomotic (Hepatobiliary disorders) | 17 | 7
Ischemic Cholangiopathy (Hepatobiliary disorders) | 2 | 1
Biliary Other (Hepatobiliary disorders) | 3 | 2
Hepatic Artery Thrombosis (Hepatobiliary disorders) | 4 | 1
Hepatic Artery Stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic Artery Other (Hepatobiliary disorders) | 1 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 1
Graft Dysfunction (Hepatobiliary disorders) | 14 | 6
Rejection (Hepatobiliary disorders) | 8 | 16
Cholangitis (Hepatobiliary disorders) | 5 | 2
Hepatic Other (Hepatobiliary disorders) | 4 | 3
Allery - Drug (Immune system disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 5 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 1
Hypertension (Cardiac disorders) | 2 | 0
Hypotension (Cardiac disorders) | 2 | 4
Hypovolemia (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 2 | 5
Tachycardia (Cardiac disorders) | 3 | 1
Arrhythmias (Cardiac disorders) | 3 | 2
Cardiovascular Other (Cardiac disorders) | 5 | 5
Hematoma/Bruising (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatologic Other (Skin and subcutaneous tissue disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 8 | 1
GI Bleed (Gastrointestinal disorders) | 5 | 3
Gastrointestinal Other (Gastrointestinal disorders) | 6 | 4
Renal Dysfunction/Acute Kidney Injury (Renal and urinary disorders) | 11 | 15
Oliguria (Renal and urinary disorders) | 1 | 0
Genitourinary Other (Renal and urinary disorders) | 5 | 0
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Other (Musculoskeletal and connective tissue disorders) | 8 | 7
Cold/Flu (Respiratory, thoracic and mediastinal disorders) | 1 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Respiratory Other (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Bleeding - No Transfusion Required (General disorders) | 2 | 0
Bleeding - Transfusion Required (General disorders) | 8 | 12
Bleeding from Hepatic Artery (General disorders) | 1 | 1
Bleeding from IVC (General disorders) | 1 | 1
Bleeding Requiring Reoperation (General disorders) | 3 | 11
Bleeding Other (General disorders) | 1 | 1
Abdominal Collection (General disorders) | 2 | 2
Pleural Effusion (General disorders) | 2 | 3
Ascites (General disorders) | 4 | 2
Extremities Edema (General disorders) | 2 | 1
Fluid Collection Other (General disorders) | 1 | 2
Pain (General disorders) | 2 | 6
Surgery - Planned/Elective (General disorders) | 5 | 4
Surgery - Emergency (General disorders) | 3 | 2
Other Systemic Disease/Event (General disorders) | 9 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 6
Leukopenia (Blood and lymphatic system disorders) | 3 | 5
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Malignancy (Blood and lymphatic system disorders) | 1 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Hematology Other (Blood and lymphatic system disorders) | 3 | 1
Hyperglycemia (Endocrine disorders) | 0 | 3
Hyperkalemia (General disorders) | 3 | 8
Hypernatremia (General disorders) | 0 | 1
Hyponatremia (General disorders) | 0 | 1
Altered Mental Status (Psychiatric disorders) | 4 | 3
Encephalopathy (Nervous system disorders) | 0 | 1
Psychiatric Disorder (Psychiatric disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 3
Stroke/TIA (Nervous system disorders) | 3 | 0
Neurology/Psychiatry Other (Psychiatric disorders) | 1 | 0
EAD - Serum Bilirubin (Hepatobiliary disorders) | 1 | 0
EAD - ALT or AST (Hepatobiliary disorders) | 5 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normothermic Machine Perfusion (NMP) (N=136) | Standard of Care (Ice) (N=131)
Hyperglycemia (Endocrine disorders) | 64 | 68
Leukopenia (Blood and lymphatic system disorders) | 33 | 28
Anemia (Blood and lymphatic system disorders) | 26 | 34
Hematology Other (Blood and lymphatic system disorders) | 9 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 9
Diarrhea (Gastrointestinal disorders) | 24 | 28
Constipation (Gastrointestinal disorders) | 25 | 26
Nausea/Vomiting (Gastrointestinal disorders) | 18 | 20
Gastrointestinal Other (Gastrointestinal disorders) | 19 | 18
Tremors (Nervous system disorders) | 21 | 19
Headache (Nervous system disorders) | 17 | 15
Altered Mental Status (Psychiatric disorders) | 15 | 9
Insomnia (Nervous system disorders) | 9 | 13
Renal Dysfunction/Acute Kidney Injury (Renal and urinary disorders) | 37 | 41
Genitourinary Other (Renal and urinary disorders) | 5 | 10
Urinary Retention (Renal and urinary disorders) | 6 | 9
UTI (Renal and urinary disorders) | 7 | 7
Hypertension (Cardiac disorders) | 25 | 25
Hypotension (Cardiac disorders) | 12 | 18
Tachycardia (Cardiac disorders) | 10 | 9
Hypovolemia (Cardiac disorders) | 7 | 7
Hypomagnesemia (General disorders) | 24 | 26
Hyperkalemia (General disorders) | 18 | 24
Hypokalemia (General disorders) | 4 | 12
Extremities Edema (General disorders) | 29 | 28
Pleural Effusion (General disorders) | 11 | 10
Graft Dysfunction (Hepatobiliary disorders) | 15 | 18
Rejection (Hepatobiliary disorders) | 11 | 7
Blood Infection (Infections and infestations) | 16 | 12
Infection Other (Infections and infestations) | 10 | 15
Other Systemic Disease/Event (General disorders) | 18 | 29
Pain (General disorders) | 14 | 15
Musculoskeletal Other (Musculoskeletal and connective tissue disorders) | 32 | 27
Respiratory Other (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Dermatologic Other (Skin and subcutaneous tissue disorders) | 15 | 17
EAD - ALT or AST (Hepatobiliary disorders) | 16 | 17
Bleeding - Transfusion Required (General disorders) | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT02775162/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT02775162/SAP_001.pdf